CLINICAL TRIAL: NCT05193851
Title: A Phase I Clinical Study Evaluating the Safety and Pharmacokinetics of Ricolinostat in Chinese Subjects
Brief Title: Evaluate the Safety and Pharmacokinetics of Ricolinostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing 3E-Regenacy Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BCRG-CN-102
Record Dates: First submitted 2021-12-08; First posted 2022-01-18 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2021-12

CONDITIONS: Peripheral Nervous System Diseases
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — ricolinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental): 12 healthy Chinese adult subjects, both male and female, are treated with ricolinostat
  Interventions: Drug: ricolinostat

INTERVENTIONS:
Drug: ricolinostat — This study is an open-label, single-dose phase I clinical study to evaluate the safety and pharmacokinetics of ricolinostat in healthy Chinese adult subjects.
  12 subjects are planned to be enrolled, both male and female, and all will receive the investigational drug.
  This study includes the screening period, baseline period, dosing/observation period, discharge and follow-up period.

SUMMARY:
This study is an open-label, phase I clinical study to evaluate the safety and pharmacokinetics of ricolinostat in healthy Chinese adult subjects.

DETAILED DESCRIPTION:
This study is an open-label, phase I clinical study to evaluate the safety and pharmacokinetics of ricolinostat in healthy Chinese adult subjects.

12 subjects are planned to be enrolled, both male and female, and all will receive the investigational drug.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who meet all of the following inclusion criteria can be enrolled in this study:

  1. Healthy adult male or female subjects aged 18 to 55 years;
  2. Body mass index of 19 - 26 kg/m2 (including the boundary value); the weight of male subjects should not be lower than 50 kg, and the weight of female subjects should not be lower than 45 kg;
  3. Subjects have no pregnancy plan and voluntarily take effective contraceptive measures during the study to 3 months after the last dose and have no sperm or egg donation plan.
  4. Subjects who fully understand the objective, nature, method and possible adverse reactions of the study, volunteer to be subjects and sign the informed consent form;
  5. Able to complete the study according to the protocol requirements.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are excluded:

  1. Allergic to ricolinostat (including excipients) and other similar drugs;
  2. Have had a history of drug abuse in the past five years or have used drugs three months before screening, or who have positive result for drug abuse screening at screening;
  3. Smokers (people who smoked tobacco products in the past 3 months), or habitual use of nicotine-containing products, or those who are tested positive for nicotine at screening;
  4. Drinking more than 14 units of alcohol per week within 6 months before screening (1 unit of alcohol = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) or have taken alcoholic products 48 hours before dosing, or tested positive for alcohol breath test;
  5. Diseases or factors judged by the investigator to be abnormal and clinically significant, including but not limited to neurological, mental, cardiovascular, blood, liver, kidney, gastrointestinal, respiratory, metabolic, endocrine, immune, skeletal system diseases or other factors;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
safety of dosed subjects | about one week
  monitor AEs

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Principal Investigator — China
Locations (1):
- Bethune First Hospital Of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No